CLINICAL TRIAL: NCT00708708
Title: A Prospective Non-interventional Study (Nis) Of The Routine Use Of Etanercept In The Long-term Treatment Of Patients With Plaque-type Psoriasis In Everyday Practice: An Efficacy, Safety, And Health Economic Evaluation
Brief Title: Observational Study Evaluating Etanercept (Enbrel®) In Subjects With Plaque-Type Psoriasis In Usual Care Settings
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881X1-4499; B1801081 (Other: Alias Study Number)
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Psoriasis
Keywords: Plaque-type psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients with moderate to severe plaque psoriasis
  Interventions: Drug: etanercept (Enbrel®)

INTERVENTIONS:
Drug: etanercept (Enbrel®) — The patients will be treated in accordance with the requirements of the labeling of etanercept in Germany. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.

SUMMARY:
This prospective observational cohort study will assess the average duration of the drug free interval between etanercept treatment cycles in usual care settings in Germany.

DETAILED DESCRIPTION:
Non-interventional study: subjects to be selected according to the usual clinical practice of their physician

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe plaque psoriasis on etanercept treatment according to the Summary of Product Characteristics (SmPC), and applicable local guidelines
* Subjects for whom the decision has already been made to initiate treatment with etanercept

Exclusion Criteria:

* Sepsis or risk of sepsis
* Current or recent infections, including chronic or localized, e.g. tuberculosis (TB) infection
* Vaccination with live vaccine in last 4 weeks, or expected to require such vaccination during the course of the study
* Pre-existing or recent onset CNS demyelinating disease.
* Class III or IV congestive heart failure as defined by the New York Heart Association classification or uncompensated congestive heart failure.
* Previous or ongoing treatment with etanercept
* Participation in other clinical or observational studies.
* Patients with psoriatic arthritis requiring continuous etanercept treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe plaque psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 926 (Actual)
Dates: Start 2008-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Westfaelische Wilhelms-Universitaet Muenster, Zentr. f. Derm, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Luger T, Schopf RE, Schwanke A, Langhammer S, Meng T, Loschmann PA. An observational study to evaluate the long-term outcomes of treatment with etanercept in patients with plaque-type psoriasis. J Eur Acad Dermatol Venereol. 2016 Oct;30(10):1730-1741. doi: 10.1111/jdv.13673. Epub 2016 Jun 14. PMID 27297981
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881X1-4499&StudyName=Observational%20Study%20Evaluating%20etanercept%20%28Enbrel%AE%29%20In%20Subjects%20With%20Plaque-Type%20Psoriasis%20In%20Usual%20Care%20Settings

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 955 participants were enrolled for documentation. Of these 955 participants enrolled, only 926 participants were included in analysis.
Groups:
- Etanercept: Participants who had moderate to severe plaque psoriasis and commenced treatment with etanercept (Enbrel) as a systemic monotherapy for the first time, received Enbrel in cycles of 24 weeks duration separated by drug-free intervals based on treating physician's discretion as per Summary of Product Characteristics (SmPC). Treatment was resumed if plaque psoriasis worsened. According to SmPC, recommended dose included etanercept 25 milligram (mg) twice weekly, 50 mg once weekly or 50 mg twice weekly subcutaneous injection. Participants were observed for 60 months.
Period: Overall Study
Arm/Group | Etanercept
Started | 955
Completed | 213 (Included participants completed total observation period and participants with planned study end.)
Not Completed | 742
Not completed — Another therapy instead of Enbrel | 141
Not completed — Lost to Follow-up | 52
Not completed — Withdrawal by Subject | 51
Not completed — Intolerance | 42
Not completed — Another therapy along with Enbrel | 15
Not completed — Other unspecified | 11
Not completed — Good effectiveness | 9
Not completed — Ineffectiveness (no systemic therapy) | 9
Not completed — Administrative reasons | 7
Not completed — Lack of effectiveness | 4
Not completed — Lack of compliance | 3
Not completed — Pregnancy | 3
Not completed — Adverse Event | 3
Not completed — Missing values | 392

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants with available post-baseline safety data.
Arm/Group | Etanercept
Number analyzed (Participants) | 926
Age, Continuous [Mean (Standard Deviation); unit: years] — Only 915 participants had data available for age.
  years | 47.4 (12.9)
Sex/Gender, Customized [Number; unit: participants]
  Female | 339
  Male | 583
  Missing values | 4

OUTCOME MEASURES:

1. Primary Outcome: Duration of Drug-Free Interval Prior to Treatment Cycle 2
Description: Average duration of participant's drug-free interval between the end of treatment Cycle 1 and Cycle 2 was reported in weeks. Duration of drug-free interval was computed as: (date of start of new treatment cycle minus date of last application of etanercept prior to drug free interval plus 1) divided by 7 and it was determined for only those participants who had information available regarding drug-free interval.
Time Frame: Cycle 1 Week 24 up to Cycle 2 Week 0
Population: Efficacy analysis set: all participants greater than or equal to (>=) 18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here 'N' (number of participants analyzed)= participants evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 120
weeks | 12.6 [10.2 to 15.0]

2. Primary Outcome: Duration of Drug-Free Interval Prior to Treatment Cycle 3
Description: Average duration of participant's drug-free interval between the end of treatment Cycle 2 and Cycle 3 was reported in weeks. Duration of drug-free interval was computed as: (date of start of new treatment cycle minus date of last application of etanercept prior to drug free interval plus 1) divided by 7 and it was determined for only those participants who had information available regarding drug-free interval.
Time Frame: Cycle 2 Week 24 up to Cycle 3 Week 0
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post-baseline documentations. Here 'N' (number of participants analyzed)= participants evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 39
weeks | 10.5 [8.2 to 12.9]

3. Primary Outcome: Duration of Drug-Free Interval Prior to Treatment Cycle 4
Description: Average duration of participant's drug-free interval between the end of treatment Cycle 3 and Cycle 4 was reported in weeks. Duration of drug-free interval was computed as: (date of start of new treatment cycle minus date of last application of etanercept prior to drug free interval plus 1) divided by 7 and it was determined for only those participants who had information available regarding drug-free interval.
Time Frame: Cycle 3 Week 24 up to Cycle 4 Week 0
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here 'N' (number of participants analyzed) = participants evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 9
weeks | 25.0 [11.7 to 38.3]

4. Primary Outcome: Duration of Drug-Free Interval Prior to Treatment Cycle 5
Description: Average duration of participant's drug-free interval between the end of treatment Cycle 4 and Cycle 5 was reported in weeks. Duration of drug-free interval was computed as: (date of start of new treatment cycle minus date of last application of etanercept prior to drug free interval plus 1) divided by 7 and it was determined for only those participants who had information available regarding drug-free interval.
Time Frame: Cycle 4 Week 24 up to Cycle 5 Week 0
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 5
weeks | 20.6 [3.9 to 37.3]

5. Primary Outcome: Duration of Drug-Free Interval Prior to Treatment Cycle 6
Description: Average duration of participant's drug-free interval between the end of treatment Cycle 5 and Cycle 6 was reported in weeks. Duration of drug-free interval was computed as: (date of start of new treatment cycle minus date of last application of etanercept prior to drug free interval plus 1) divided by 7 and it was determined for only those participants who had information available regarding drug-free interval.
Time Frame: Cycle 5 Week 24 up to Cycle 6 Week 0
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 2
weeks | 14.2 [-1.2 to 29.6]

6. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections: head, arms, trunk, legs. For each section, percent (%) area of skin involved was estimated: 0= 0% to 6= 90-100%. Severity was estimated by clinical signs: erythema, induration, desquamation; scale: 0= none to 4= maximum. Final PASI = sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4); total possible score range: 0= no disease to 72= maximal disease. PASI score at Week 0 of each cycle signifies the disease activity at the time of resumption of etanercept therapy.
Time Frame: Week 0, 12, 24 of Cycle 1 to 6
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here 'n' = participants evaluable for this measure at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 720
units on a scale
  Cycle 1 Week 0 (n=675) | 21.0 (12.1)
  Cycle 1 Week 12 (n=605) | 8.8 (8.5)
  Cycle 1 Week 24 (n=538) | 5.9 (6.6)
  Cycle 2 Week 0 (n=435) | 6.7 (6.5)
  Cycle 2 Week 12 (n=394) | 4.9 (5.0)
  Cycle 2 Week 24 (n=368) | 4.8 (5.2)
  Cycle 3 Week 0 (n=234) | 4.9 (6.1)
  Cycle 3 Week 12 (n=226) | 4.2 (5.5)
  Cycle 3 Week 24 (n=202) | 3.6 (4.5)
  Cycle 4 Week 0 (n=120) | 3.9 (3.9)
  Cycle 4 Week 12 (n=117) | 4.2 (3.6)
  Cycle 4 Week 24 (n=105) | 4.1 (4.8)
  Cycle 5-week 0 (n=77) | 3.6 (3.0)
  Cycle 5 Week 12 (n=79) | 4.2 (4.1)
  Cycle 5 Week 24 (n=63) | 3.6 (3.2)
  Cycle 6 Week 0 (n=60) | 3.9 (3.6)
  Cycle 6 Week 12 (n=54) | 3.0 (3.4)
  Cycle 6 Week 24 (n=48) | 2.8 (2.7)

7. Secondary Outcome: Percentage of Body Surface Area (BSA) Affected by Psoriasis
Description: Percentage of body surface area affected by psoriasis was estimated using the palm method: one of the participant's palm to proximal interphalangeal and thumb = 1% of total BSA. Regions of the body were assigned specific number of palms with percentage [Head and neck = 10% (10 palms), upper extremities = 20% (20 palms), Trunk (axillae and groin) = 30% (30 palms), lower extremities (buttocks) = 40% (40 palms)]. The total BSA affected was the summation of individual regions affected. The results of this outcome measure was summarized separately for participants without drug-free interval, participants with drug-free interval and remaining participants, as per planned analysis.
Time Frame: Week 0, 12, 24 of Cycle 1 to 6
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here 'n' = participants evaluable for this measure at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Groups:
- Participants Without Drug-Free Interval: Participants who had moderate to severe plaque psoriasis and commenced treatment with etanercept (Enbrel) as a systemic monotherapy for the first time, received Enbrel in cycles of 24 weeks duration separated by drug-free intervals based on treating physician's discretion as per Summary of Product Characteristics (SmPC). Treatment was resumed if plaque psoriasis worsened. According to SmPC, recommended dose included etanercept 25 mg twice weekly, 50 mg once weekly or 50 mg twice weekly subcutaneous injection. Participants were observed for 60 months. This group included participants who never experienced a drug-free interval during the entire observational period.
- Participants With Drug-Free Interval: Participants who had moderate to severe plaque psoriasis and commenced treatment with etanercept (Enbrel) as a systemic monotherapy for the first time, received Enbrel in cycles of 24 weeks duration separated by drug-free intervals based on treating physician's discretion as per Summary of Product Characteristics (SmPC). Treatment was resumed if plaque psoriasis worsened. According to SmPC, recommended dose included etanercept 25 mg twice weekly, 50 mg once weekly or 50 mg twice weekly subcutaneous injection. Participants were observed for 60 months. This group included participants who were always treated with a drug-free interval during the observational period.
- Remaining Participants: Participants who had moderate to severe plaque psoriasis and commenced treatment with etanercept (Enbrel) as a systemic monotherapy for the first time, received Enbrel in cycles of 24 weeks duration separated by drug-free intervals based on treating physician's discretion as per Summary of Product Characteristics (SmPC). Treatment was resumed if plaque psoriasis worsened. According to SmPC, recommended dose included etanercept 25 mg twice weekly, 50 mg once weekly or 50 mg twice weekly subcutaneous injection. Participants were observed for 60 months. This group included participants who experienced both, treatment with and without drug-free interval during the observational period.
Arm/Group | Participants Without Drug-Free Interval | Participants With Drug-Free Interval | Remaining Participants
Number analyzed (Participants) | 298 | 147 | 275
percentage of BSA
  Cycle 1 Week 0 (n=293,145,267) | 28.2 (20.8) | 36.7 (21.3) | 35.1 (23.2)
  Cycle 1 Week 12 (n=293,142,235) | 14.0 (13.6) | 20.1 (18.0) | 21.6 (19.8)
  Cycle 1 Week 24 (n=294,143,168) | 9.4 (10.3) | 13.6 (15.1) | 15.9 (17.6)
  Cycle 2 Week 0 (n=293,143,66) | 9.4 (10.3) | 18.7 (15.0) | 11.6 (13.1)
  Cycle 2 Week 12 (n=280,127,62) | 8.4 (9.8) | 12.6 (14.3) | 11.1 (13.4)
  Cycle 2 Week 24 (n=263,117,53) | 7.7 (9.4) | 10.3 (11.0) | 9.2 (10.1)
  Cycle 3 Week 0 (n=212,44,47) | 7.3 (9.5) | 13.9 (13.3) | 10.7 (13.0)
  Cycle 3 Week 12 (n=201,40,43) | 6.6 (8.0) | 9.9 (12.8) | 9.7 (13.5)
  Cycle 3 Week 24 (n=181,38,36) | 6.3 (7.2) | 6.8 (9.1) | 8.8 (11.0)
  Cycle 4 Week 0 (n=144,8,21) | 6.0 (6.0) | 16.5 (13.8) | 8.2 (9.8)
  Cycle 4 Week 12 (n=128,8,20) | 5.9 (5.6) | 7.9 (5.2) | 8.2 (11.4)
  Cycle 4 Week 24 (n=121,7,18) | 6.2 (6.4) | 10.3 (8.2) | 5.4 (6.6)
  Cycle 5 Week 0 (n=100,4,10) | 6.1 (5.8) | 19.8 (8.8) | 7.2 (8.1)
  Cycle 5 Week 12 (n=98,2,9) | 6.0 (6.7) | 17.5 (10.6) | 4.8 (4.5)
  Cycle 5 Week 24 (n=88,1,5) | 6.0 (7.3) | 5.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point. | 3.4 (1.5)
  Cycle 6 Week 0 (n=82,1,3) | 6.2 (7.5) | 5.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point. | 4.0 (3.5)
  Cycle 6 Week 12 (n=75,0,2) | 5.7 (6.8) | NA (NA) — Data was not reported since no participant was evaluable at this time point. | 3.0 (1.4)
  Cycle 6 Week 24 (n=68,0,2) | 5.2 (7.4) | NA (NA) — Data was not reported since no participant was evaluable at this time point. | 2.0 (0.0)

8. Secondary Outcome: Static Physician Global Assessment (sPGA) of Disease Activity
Description: Static physician global assessment (sPGA) of disease activity was assessed as 0 (no psoriasis) to 5 (severe disease) based on severity of induration, scaling, and erythema across all psoriatic lesions.
Time Frame: Week 0, 12, 24 of Cycle 1 to 6
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. 'n'= participants evaluable for this measure at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 720
units on a scale
  Cycle 1 Week 0 (n=718) | 3.1 (0.9)
  Cycle 1 Week 12 (n=683) | 1.9 (1.0)
  Cycle 1 Week 24 (n=615) | 1.6 (1.0)
  Cycle 2 Week 0 (n=514) | 1.7 (1.0)
  Cycle 2 Week 12 (n=482) | 1.5 (0.9)
  Cycle 2 Week 24 (n=444) | 1.5 (1.0)
  Cycle 3 Week 0 (n=307) | 1.5 (1.0)
  Cycle 3 Week 12 (n=291) | 1.4 (1.0)
  Cycle 3 Week 24 (n=259) | 1.3 (0.9)
  Cycle 4 Week 0 (n=174) | 1.4 (0.9)
  Cycle 4 Week 12 (n=158) | 1.5 (0.9)
  Cycle 4 Week 24 (n=147) | 1.5 (0.9)
  Cycle 5 Week 0 (n=114) | 1.5 (0.8)
  Cycle 5 Week 12 (n=109) | 1.6 (0.9)
  Cycle 5 Week 24 (n=95) | 1.5 (0.8)
  Cycle 6 Week 0 (n=88) | 1.5 (0.9)
  Cycle 6 Week 12 (n=78) | 1.3 (0.8)
  Cycle 6 Week 24 (n=71) | 1.3 (0.8)

9. Secondary Outcome: Physician Global Assessment of Efficacy
Description: Physician assessed the effectiveness of etanercept treatment at the end (Week 24) of each cycle as very good, good, moderate, and insufficient.
Time Frame: Week 24 of Cycle 1 to 6
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here 'n'= number of participants evaluable at the end of the given cycles for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 720
participants
  Cycle 1: very good (n=606) | 304 (0.9)
  Cycle 1: good (n=606) | 214 (1.0)
  Cycle 1: moderate (n=606) | 68 (1.0)
  Cycle 1: insufficient (n=606) | 20 (1.0)
  Cycle 2: very good (n=440) | 242 (0.9)
  Cycle 2: good (n=440) | 151 (1.0)
  Cycle 2: moderate (n=440) | 39 (1.0)
  Cycle 2: insufficient (n=440) | 8 (1.0)
  Cycle 3: very good (n=259) | 153 (0.9)
  Cycle 3: good (n=259) | 92 (0.9)
  Cycle 3: moderate (n=259) | 13 (0.9)
  Cycle 3: insufficient (n=259) | 1 (0.9)
  Cycle 4: very good (n=147) | 81 (0.8)
  Cycle 4: good (n=147) | 59 (0.9)
  Cycle 4: moderate (n=147) | 4 (0.8)
  Cycle 4: insufficient (n=147) | 3 (0.9)
  Cycle 5: very good (n=96) | 53 (0.8)
  Cycle 5: good (n=96) | 40 (0.8)
  Cycle 5: moderate (n=96) | 3
  Cycle 5: insufficient (n=96) | 0
  Cycle 6: very good (n=70) | 49
  Cycle 6: good (n=70) | 18
  Cycle 6: moderate (n=70) | 3
  Cycle 6: insufficient (n=70) | 0

10. Secondary Outcome: Patient Global Assessment of Efficacy
Description: Participant assessed the effectiveness of etanercept treatment at the end (Week 24) of each cycle as very good, good, moderate, and insufficient.
Time Frame: Week 24 of Cycle 1 to 6
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 720
participants
  Cycle 1: very good (n=605) | 297 (0.9)
  Cycle 1: good (n=605) | 216 (1.0)
  Cycle 1: moderate (n=605) | 65 (1.0)
  Cycle 1: insufficient (n=605) | 27 (1.0)
  Cycle 2: very good (n=444) | 229 (0.9)
  Cycle 2: good (n=444) | 165 (1.0)
  Cycle 2: moderate (n=444) | 40 (1.0)
  Cycle 2: insufficient (n=444) | 10 (1.0)
  Cycle 3: very good (n=258) | 145 (0.9)
  Cycle 3: good (n=258) | 98 (0.9)
  Cycle 3: moderate (n=258) | 10 (0.9)
  Cycle 3: insufficient (n=258) | 5 (0.9)
  Cycle 4: very good (n=147) | 77 (0.8)
  Cycle 4: good (n=147) | 61 (0.9)
  Cycle 4: moderate (n=147) | 7 (0.8)
  Cycle 4: insufficient (n=147) | 2 (0.9)
  Cycle 5: very good (n=96) | 39 (0.8)
  Cycle 5: good (n=96) | 50 (0.8)
  Cycle 5: moderate (n=96) | 7
  Cycle 5: insufficient (n=96) | 0
  Cycle 6: very good (n=71) | 47
  Cycle 6: good (n=71) | 21
  Cycle 6: moderate (n=71) | 3
  Cycle 6: insufficient (n=71) | 0

11. Secondary Outcome: Number of Injections Per Year
Description: Number of etanercept injections per year were calculated up to 5 years. 'By year' analysis was not possible for those participants for whom the data of one or more visits was missing.
Time Frame: Year 1, 2, 3, 4, 5
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. 'n'= participants evaluable at the specified time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Etanercept
Number analyzed (Participants) | 720
injections
  Year 1 (n=675) | 47.0 (22.2)
  Year 2 (n=418) | 30.8 (22.4)
  Year 3 (n=167) | 32.1 (20.3)
  Year 4 (n=53) | 15.6 (12.9)
  Year 5 (n=7) | 11.8 (10.3)

12. Secondary Outcome: Cumulative Dose of Etanercept Per Year
Description: Cumulative dose of etanercept per year was calculated up to 5 years. 'By year' analysis was not possible for those participants for whom the data of one or more visits was missing.
Time Frame: Year 1, 2, 3, 4, 5
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. 'n' = participants evaluable at the specified time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Etanercept
Number analyzed (Participants) | 720
mg
  Year 1 (n=664) | 2249.2 (1100.6)
  Year 2 (n=418) | 1474.7 (1104.6)
  Year 3 (n=167) | 1565.5 (1027.3)
  Year 4 (n=53) | 729.1 (589.9)
  Year 5 (n=7) | 399.5 (354.5)

13. Secondary Outcome: Percentage of Time on Treatment in First Year
Description: Percentage of time on etanercept treatment for first year was calculated. It was calculated as 100% * (365- sum of durations of drug-free intervals in the first year)/365. Analysis was not possible for participants with missing data of visit 1 (Week 0) of Cycle 1.
Time Frame: Year 1
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: percentage of first year
Arm/Group | Etanercept
Number analyzed (Participants) | 677
percentage of first year | 96.5 (10.6)

14. Secondary Outcome: Percentage of Time on Treatment Over Entire Period
Description: Percentage of time on etanercept treatment over entire treatment period was calculated. It was calculated as 100% * ([Date of last application - Date of first application + 1] - Sum of duration of drug-free intervals [days])/(Date of last application - Date of first application + 1).
Time Frame: Cycle 1 up to Cycle 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of entire treatment period
Arm/Group | Etanercept
Number analyzed (Participants) | 400
percentage of entire treatment period | 94.8 (10.9)

15. Secondary Outcome: Patient's Global Assessment of Disease Activity (PatGA)
Description: Participants were asked to rate the severity of their disease activity on a 6-point scale, where 0 = no activity and 5 = severe or maximum activity.
Time Frame: Week 0, 12, 24 of Cycle 1 to 6
Population: Efficacy analysis set included all participants >=18 years of age, confirmed diagnosis of plaque psoriasis, had not received treatment with etanercept previously and had post baseline documentations. Here, 'n'=number of participants evaluable for this measure at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 720
units on a scale
  Cycle 1 Week 0 (n=673) | 3.7 (1.2)
  Cycle 1 Week 12 (n=629) | 2.2 (1.2)
  Cycle 1 Week 24 (n=554) | 1.9 (1.2)
  Cycle 2 Week 0 (n=349) | 2.2 (1.3)
  Cycle 2 Week 12 (n=455) | 1.7 (1.1)
  Cycle 2 Week 24 (n=395) | 1.7 (1.2)
  Cycle 3 Week 0 (n=191) | 1.8 (1.2)
  Cycle 3 Week 12 (n=261) | 1.6 (1.1)
  Cycle 3 Week 24 (n=224) | 1.6 (1.2)
  Cycle 4 Week 0 (n=89) | 1.8 (1.1)
  Cycle 4 Week 12 (n=145) | 1.7 (1.1)
  Cycle 4 Week 24 (n=132) | 1.8 (1.1)
  Cycle 5 Week 0 (n=63) | 1.9 (1.1)
  Cycle 5 Week 12 (n=103) | 1.7 (1.0)
  Cycle 5 Week 24 (n=92) | 1.8 (0.9)
  Cycle 6 Week 0 (n=43) | 2.2 (0.9)
  Cycle 6 Week 12 (n=76) | 1.6 (1.1)
  Cycle 6 Week 24 (n=68) | 1.6 (1.0)

16. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score
Description: DLQI is the dermatology-specific quality of life measure used for psoriatic population. The 10-item questionnaire has a score range of 0 to 30 with higher scores indicating poor quality of life. An estimate of the minimal clinically important difference of the DLQI total score is a 5 point improvement. Total score range: 0 (best) to 30 (worst).
Time Frame: Week 0, 12, 24 of Cycle 1 to 6
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here, 'n'=number of participants evaluable for this measure at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 720
units on a scale
  Cycle 1 Week 0 (n=654) | 14.0 (7.3)
  Cycle 1 Week 12 (n=598) | 6.4 (5.8)
  Cycle 1 Week 24 (n=536) | 4.9 (5.7)
  Cycle 2 Week 0 (n=334) | 6.2 (6.3)
  Cycle 2 Week 12 (n=440) | 4.3 (5.1)
  Cycle 2 Week 24 (n=378) | 4.2 (5.3)
  Cycle 3 Week 0 (n=186) | 4.9 (5.9)
  Cycle 3 Week 12 (n= 258) | 3.9 (5.1)
  Cycle 3 Week 24 (n=221) | 3.7 (5.0)
  Cycle 4 Week 0 (n=90) | 4.7 (6.4)
  Cycle 4 Week 12 (n=146) | 3.6 (4.4)
  Cycle 4 Week 24 (n=132) | 3.8 (5.1)
  Cycle 5 Week 0 (n=64) | 4.5 (5.4)
  Cycle 5 Week 12 (n=104) | 3.8 (4.8)
  Cycle 5 Week 24 (n=91) | 3.7 (4.3)
  Cycle 6 Week 0 (n=43) | 5.0 (5.1)
  Cycle 6 Week 12 (n=75) | 3.5 (4.6)
  Cycle 6 Week 24 (n=69) | 3.9 (4.4)

17. Secondary Outcome: Euro Quality of Life-5 Dimensions (EQ-5D) Time Trade Off (TTO)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (extreme problems). Score of each domain is transformed into a single TTO value using formula developed by Greiner et al and results in a total score range -0.205 to 0.999; higher score indicates a better health state.
Time Frame: Week 0, 12, 24 of Cycle 1 to 6
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 720
units on a scale
  Cycle 1 Week 0 (n=666 ) | 0.817 (0.236)
  Cycle 1 Week 12 (n=628) | 0.915 (0.149)
  Cycle 1 Week 24 (n=549) | 0.930 (0.145)
  Cycle 2 Week 0 (n=344) | 0.915 (0.154)
  Cycle 2 Week 12 (n=451) | 0.933 (0.142)
  Cycle 2 Week 24 (n=393) | 0.939 (0.140)
  Cycle 3 Week 0 (n=190) | 0.932 (0.149)
  Cycle 3 Week 12 (n= 257) | 0.949 (0.094)
  Cycle 3 Week 24 (n=222) | 0.928 (0.154)
  Cycle 4 Week 0 (n=89) | 0.912 (0.169)
  Cycle 4 Week 12 (n=144) | 0.935 (0.121)
  Cycle 4 Week 24 (n=129) | 0.927 (0.153)
  Cycle 5 Week 0 (n=63) | 0.914 (0.157)
  Cycle 5 Week 12 (n=104) | 0.932 (0.103)
  Cycle 5 Week 24 (n=91) | 0.950 (0.099)
  Cycle 6 Week 0 (n=43) | 0.930 (0.097)
  Cycle 6 Week 12 (n=75) | 0.938 (0.098)
  Cycle 6 Week 24 (n=69) | 0.939 (0.127)

18. Secondary Outcome: Euro Quality of Life (EQ-5D)- Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state. Score of each domain is transformed into a single VAS score using formula developed by Greiner et al and results in a total score range of 0 to 100, where higher score indicates a better health state.
Time Frame: Week 0, 12, 24 of Cycle 1 to 6
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 720
units on a scale
  Cycle 1 Week 0 (n=666 ) | 73.8 (20.5)
  Cycle 1 Week 12 (n=628) | 85.1 (16.7)
  Cycle 1 Week 24 (n=549) | 87.7 (16.9)
  Cycle 2 Week 0 (n=344) | 85.6 (17.7)
  Cycle 2 Week 12 (n=451) | 88.6 (15.9)
  Cycle 2 Week 24 (n=393) | 89.5 (16.3)
  Cycle 3 Week 0 (n=190) | 88.3 (17.0)
  Cycle 3 Week 12 (n= 257) | 90.3 (14.0)
  Cycle 3 Week 24 (n=222) | 88.5 (17.7)
  Cycle 4 Week 0 (n=89) | 85.7 (18.9)
  Cycle 4 Week 12 (n=144) | 88.8 (15.4)
  Cycle 4 Week 24 (n=129) | 87.8 (17.9)
  Cycle 5 Week 0 (n=63) | 85.0 (18.8)
  Cycle 5 Week 12 (n=104) | 87.1 (15.4)
  Cycle 5 Week 24 (n=91) | 89.4 (14.9)
  Cycle 6 Week 0 (n=43) | 85.1 (16.2)
  Cycle 6 Week 12 (n=75) | 87.8 (13.8)
  Cycle 6 Week 24 (n=69) | 89.0 (14.9)

19. Secondary Outcome: Number of Participants With at Least 1 Concomitant Medication
Description: Number of participants taking any non-study medications which were administered during the period of etanercept treatment for the management of an adverse event or for the treatment of any other disease and not plaque psoriasis were reported.
Time Frame: Cycle 1 Week 0 up to Cycle 6 Week 24
Population: Safety analysis set included all participants with available post-baseline safety data.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 926
participants | 368 (10.6)

20. Secondary Outcome: Annual Costs for Treatment With Etanercept
Description: Costs for treatment with etanercept per year up to 5 years was calculated in Euros. 'By year' analysis was not possible for those participants for whom the data of 1 or more visits was missing.
Time Frame: Year 1, 2, 3, 4, 5
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here 'n'= participants evaluable at the specified time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: Euros
Arm/Group | Etanercept
Number analyzed (Participants) | 720
Euros
  Year 1 (n=675) | 20670.0 (9743.9)
  Year 2 (n=418) | 13509.6 (9854.3)
  Year 3 (n=167) | 14113.4 (8913.8)
  Year 4 (n=53) | 6847.4 (5648.6)
  Year 5 (n=7) | 5173.7 (4506.6)

21. Secondary Outcome: Average Cost of Treatment by Disease Severity
Description: Average costs for treatment with etanercept up to 5 years was calculated in Euros. Disease severity was categorized as mild (0 to 10 PASI score), moderate (10.1 to 20 PASI score) and severe (20.1 to 72 PASI score) at each year. PASI: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections: head, arms, trunk, legs. For each section, percent area of skin involved was estimated: 0= 0% to 6= 90-100%. Severity was estimated by clinical signs: erythema, induration, desquamation; scale: 0= none to 4= maximum. Final PASI = sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4); total possible score range: 0= no disease to 72= maximal disease. 'By year' analysis was not possible for those participants for whom the data of one or more visits was missing.
Time Frame: Year 1, 2, 3, 4, 5
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here 'n'= participants evaluable at the specified time points for the given disease severities.
Measure: Mean (Standard Deviation); unit: Euros
Arm/Group | Etanercept
Number analyzed (Participants) | 720
Euros
  Year 1: Mild (n=290) | 20707.0 (9751.6)
  Year 1: Moderate (n=80) | 21627.0 (11119.5)
  Year 1: Severe (n=46) | 21309.2 (11573.3)
  Year 2: Mild (n=200) | 13777.1 (9864.5)
  Year 2: Moderate (n=32) | 9668.8 (7638.6)
  Year 2: Severe (n=9) | 5479.7 (4225.8)
  Year 3: Mild (n=93) | 15062.1 (8676.5)
  Year 3: Moderate (n=3) | 6877.2 (3071.3)
  Year 3: Severe (n=4) | 6371.3 (2565.0)
  Year 4: Mild (n=25) | 5809.6 (3125.3)
  Year 4: Moderate (n=1) | 7467.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Year 4: Severe (n=2) | 3196.0 (575.5)
  Year 5: Mild (n=6) | 5309.3 (4998.2)

22. Secondary Outcome: Amount of Annual Cost for Participants Arising From Out-of-Pocket Payment and Concomitant Medications
Description: Annual costs for participants for treatment with etanercept due to out of pocket payments (included payments which were not reimbursed by the health insurance funds) and concomitant medications was reported per month for costs prior to study and per year for each year in the study up to 5 years. 'By year' analysis was not possible for those participants for whom the data of 1 or more visits was missing.
Time Frame: Prior to study, Year 1, 2, 3, 4, 5
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Euros
Arm/Group | Etanercept
Number analyzed (Participants) | 720
Euros
  Prior to Study (n=536) | 77.1 (170.6)
  Year 1 (n=472) | 194.8 (729.3)
  Year 2 (n=312) | 91.2 (445.7)
  Year 3 (n=131) | 128.8 (956.9)
  Year 4 (n=44) | 31.5 (87.6)
  Year 5 (n=6) | 53.6 (49.9)

23. Secondary Outcome: Effect of Drug-Free Interval on Patient's Global Assessment of Disease Activity (PatGA)
Description: Effect of drug-free interval on PatGA was determined by comparing the PatGA scores of the sub group "Participants Without Drug-Free Interval" to that of the sub group "Participants With Drug-Free Interval". PatGA: participants were asked to rate the severity of their disease activity on a 6-point scale, where 0 = no activity and 5 = severe or maximum activity.
Time Frame: Week 0, 12, 24 of Cycle 1 to 6
Population: Efficacy analysis set: all participants >=18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here, 'n'=number of participants evaluable for this measure at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Without Drug-Free Interval | Participants With Drug-Free Interval
Number analyzed (Participants) | 298 | 147
units on a scale
  Cycle 1 Week 0 (n=280, 138) | 3.7 (1.2) | 3.9 (0.9)
  Cycle 1 Week 12 (n=279, 138) | 2.1 (1.2) | 2.1 (1.3)
  Cycle 1 Week 24 (n=274, 139) | 1.9 (1.1) | 1.8 (1.3)
  Cycle 2 Week 0 (n=156, 136) | 2.0 (1.2) | 2.6 (1.3)
  Cycle 2 Week 12 (n=264, 130) | 1.8 (1.2) | 1.8 (1.0)
  Cycle 2 Week 24 (n=238, 111) | 1.7 (1.2) | 1.7 (1.3)
  Cycle 3 Week 0 (n=112, 41) | 1.8 (1.2) | 2.1 (1.3)
  Cycle 3 Week 12 (n=184, 38) | 1.7 (1.2) | 1.5 (1.1)
  Cycle 3 Week 24 (n=161, 36) | 1.7 (1.2) | 1.2 (1.2)
  Cycle 4 Week 0 (n=71, 6) | 1.8 (1.1) | 2.2 (1.5)
  Cycle 4 Week 12 (n=123, 6) | 1.7 (1.1) | 2.0 (1.3)
  Cycle 4 Week 24 (n=112, 5) | 1.8 (1.0) | 3.2 (1.8)
  Cycle 5 Week 0 (n=53, 2) | 1.9 (1.1) | 3.0 (1.4)
  Cycle 5 Week 12 (n=94, 2) | 1.6 (1.0) | 3.0 (1.4)
  Cycle 5 Week 24 (n=84, 2) | 1.8 (0.9) | 3.0 (1.4)
  Cycle 6 Week 0 (n=39, 2) | 2.2 (0.8) | 3.5 (0.7)
  Cycle 6 Week 12 (n=73 1) | 1.6 (1.1) | 3.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Cycle 6 Week 24(n=66, 0) | 1.7 (1.0) | NA (NA) — Data was not reported since no participant was evaluable at this time point.

24. Secondary Outcome: Effect of Drug-Free Interval on Dermatology Life Quality Index (DLQI) Score
Description: Effect of drug free interval on DLQI was determined by comparing the scores of the sub group "Participants Without Drug-Free Interval" to that of the sub group "Participants With Drug-Free Interval". DLQI is the dermatology-specific quality of life measure used for psoriatic population. The 10-item questionnaire has a score range of 0 to 30 with higher scores indicating poor quality of life. An estimate of the minimal clinically important difference of the DLQI total score is a 5 point improvement. Total score range: 0 (best) to 30 (worst).
Time Frame: Week 0, 12, 24 of Cycle 1 to 6
Population: Efficacy analysis set: all participants >= 18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here 'n'=number of participants evaluable at the specified time points for the given cycles.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Without Drug-Free Interval | Participants With Drug-Free Interval
Number analyzed (Participants) | 298 | 147
units on a scale
  Cycle 1 Week 0 (n=276,136) | 13.8 (7.3) | 15.5 (7.2)
  Cycle 1 Week 12 (n=267,126) | 5.7 (5.3) | 7.1 (5.9)
  Cycle 1 Week 24 (n=263,135) | 4.7 (5.6) | 4.7 (5.5)
  Cycle 2 Week 0 (n=145,133) | 5.8 (6.4) | 7.6 (6.5)
  Cycle 2 Week 12 (n=256,128) | 4.4 (5.4) | 4.5 (4.9)
  Cycle 2 Week 24 (n=227,107) | 4.4 (5.8) | 4.0 (4.4)
  Cycle 3 Week 0 (n=109,41) | 5.0 (6.2) | 6.4 (6.5)
  Cycle 3 Week 12 (n= 183,38) | 4.2 (5.4) | 3.7 (5.0)
  Cycle 3 Week 24 (n=158,36) | 4.1 (5.5) | 2.1 (3.0)
  Cycle 4 Week 0 (n=72,6) | 5.0 (6.4) | 4.5 (9.1)
  Cycle 4 Week 12 (n=124,6) | 3.6 (4.5) | 4.5 (5.5)
  Cycle 4 Week 24 (n=112,5) | 3.9 (5.2) | 5.0 (5.7)
  Cycle 5 Week 0 (n=53,3) | 4.8 (5.8) | 1.7 (1.5)
  Cycle 5 Week 12 (n=94,2) | 3.7 (4.7) | 3.0 (0.0)
  Cycle 5 Week 24 (n=83,2) | 3.7 (4.4) | 3.0 (1.4)
  Cycle 6 Week 0 (n=39,2) | 5.1 (5.3) | 5.5 (2.1)
  Cycle 6 Week 12 (n=72,1) | 3.6 (4.7) | 1.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Cycle 6 Week 24 (n=67,0) | 4.0 (4.4) | NA (NA) — Data was not reported since no participant was evaluable at this time point.

25. Secondary Outcome: Effect of Drug-Free Interval on Euro Quality of Life-5 Dimensions (EQ-5D) Time Trade-Off (TTO)
Description: Effect of drug free interval on EQ-5D was determined by comparing the scores of the sub group "Participants Without Drug-Free Interval" to that of the sub group "Participants With Drug-Free Interval". EQ-5D: participant rated questionnaire to assess health-related quality of life. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (extreme problems). Score of each domain is transformed into a single TTO value using formula developed by Greiner et al and results in a total score range -0.205 to 0.999; higher score indicates a better health state.
Time Frame: Week 0, 12, 24 of Cycle 1 to 6
Population: Efficacy analysis set: all participants >= 18 years of age, confirmed diagnosis of moderate or severe plaque psoriasis, who received etanercept monotherapy for the first time during the study and had post baseline documentations. Here n'=number of participants evaluable at the specified time points for the given cycles.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Without Drug-Free Interval | Participants With Drug-Free Interval
Number analyzed (Participants) | 298 | 147
units on a scale
  Cycle 1 Week 0 (n=279,137) | 0.810 (0.243) | 0.809 (0.232)
  Cycle 1 Week 12 (n=281,137) | 0.914 (0.144) | 0.916 (0.151)
  Cycle 1 Week 24 (n=272,139) | 0.921 (0.149) | 0.944 (0.117)
  Cycle 2 Week 0 (n=152,135) | 0.903 (0.164) | 0.920 (0.144)
  Cycle 2 Week 12 (n=261,129) | 0.930 (0.140) | 0.949 (0.128)
  Cycle 2 Week 24 (n=238,111) | 0.934 (0.148) | 0.948 (0.123)
  Cycle 3 Week 0 (n=111,41) | 0.931 (0.139) | 0.921 (0.183)
  Cycle 3 Week 12 (n= 181,37) | 0.946 (0.088) | 0.969 (0.049)
  Cycle 3 Week 24 (n=160,35) | 0.921 (0.157) | 0.972 (0.068)
  Cycle 4 Week 0 (n=71,6) | 0.894 (0.184) | 0.980 (0.046)
  Cycle 4 Week 12 (n=122,6) | 0.929 (0.129) | 0.962 (0.058)
  Cycle 4 Week 24 (n=110,5) | 0.920 (0.163) | 0.954 (0.061)
  Cycle 5 Week 0 (n=53,2) | 0.907 (0.168) | 0.943 (0.079)
  Cycle 5 Week 12 (n=94,2) | 0.929 (0.107) | 0.943 (0.079)
  Cycle 5 Week 24 (n=83,2) | 0.950 (0.101) | 0.943 (0.079)
  Cycle 6 Week 0 (n=39,2) | 0.932 (0.101) | 0.887 (0.000)
  Cycle 6 Week 12 (n=72,1) | 0.939 (0.100) | 0.887 (NA) — Standard deviation was not estimable as only 1 participant was analyzed at this time-point.
  Cycle 6 Week 24 (n=67,0) | 0.937 (0.128) | NA (NA) — Data was not reported since no participant was evaluable at this time point.

26. Secondary Outcome: Participant Perception of Drug-Free Interval: Length of Drug-Free Interval
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). Before the drug-free interval participants were asked, "How long do you expect the drug-free interval to last for?" After the drug-free interval participants were asked, "How long did the drug-free interval last?" Results are reported for participant's perception of the length of drug-free interval.
Time Frame: Before Cycle 2, 3, 4, 5, 6, after Cycle 1, 2, 3, 4, 5
Population: Efficacy analysis set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure; 'n' signifies those participants who were evaluable for this measure at the specified time points.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Etanercept
Number analyzed (Participants) | 102
months
  After Cycle 1 (n=50) | 0.9 (1.0)
  Before Cycle 2 (n=102) | 2.4 (2.9)
  After Cycle 2 (n=19) | 1.4 (1.5)
  Before Cycle 3 (n=37) | 1.6 (1.6)
  After Cycle 3 (n=2) | 4.5 (2.1)
  Before Cycle 4 (n=5) | 1.8 (1.8)
  After Cycle 4 (n=0) | NA (NA) — Mean and standard deviation were not estimable as no participant was evaluable at this time point.
  Before Cycle 5 (n=1) | 2.3 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  After Cycle 5 (n=0) | NA (NA) — Mean and standard deviation were not estimable as no participant was evaluable at this time point.
  Before Cycle 6 (n=1) | 2.8 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.

27. Secondary Outcome: Participant Perception of Drug-Free Interval: Reason for Returning to Practice
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). After the drug-free interval participants were asked, "Why did you return to the practice today?" Responses included unscheduled visit due to new occurrence of disease, scheduled visit or other reasons (included reasons like treatment of adverse event, get a prescription or examination after external treatment). Results are reported for reasons for returning to the practice.
Time Frame: Before Cycle 2, 3, 4, 5, 6
Population: Efficacy analysis set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure; 'n' signifies those participants who were evaluable for this measure at the specified time points.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 116
participants
  Before Cycle 2- unscheduled visit (n=116) | 66 (2.9)
  Before Cycle 2- scheduled visit (n=116) | 46 (1.0)
  Before Cycle 2- other reason (n=116) | 4 (1.6)
  Before Cycle 3- unscheduled visit (n=43) | 16 (1.5)
  Before Cycle 3- scheduled visit (n=43) | 26 (1.8)
  Before Cycle 3- other reason (n=43) | 1
  Before Cycle 4- unscheduled visit(n=7) | 2
  Before Cycle 4- scheduled visit (n=7) | 4
  Before Cycle 4-other reason (n=7) | 1
  Before Cycle 5- unscheduled visit(n=1) | 0
  Before Cycle 5-scheduled visit (n=1) | 1
  Before Cycle 5-other reason (n=1) | 0
  Before Cycle 6- unscheduled visit (n=1) | 0
  Before Cycle 6-scheduled visit (n=1) | 1
  Before Cycle 6-other reason (n=1) | 0

28. Secondary Outcome: Participant Perception of Drug-Free Interval: Liking of Drug-Free Interval
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). Before the drug-free interval participants were asked, "Do you basically like the idea of a drug-free interval?" After the drug-free interval participants were asked, "How did you like the current drug-free interval?" Participants responded on a scale of 1 (not at all) to 5 (very good). Results are reported for participant's liking of the drug-free interval.
Time Frame: Before Cycle 2, 3, 4, 5, 6, after Cycle 1, 2, 3, 4, 5
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 113
units on a scale
  After Cycle 1 (n=113) | 2.6 (1.5)
  Before Cycle 2 (n=106) | 2.5 (1.4)
  After Cycle 2 (n=40) | 3.1 (1.5)
  Before Cycle 3 (n=37) | 2.9 (1.4)
  After Cycle 3 (n=7) | 2.1 (1.7)
  Before Cycle 4 (n=5) | 1.0 (0.0)
  After Cycle 4 (n=2) | 1.5 (0.7)
  Before Cycle 5 (n=1) | 2.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  After Cycle 5 (n=1) | 4.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6 (n=1) | 2.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.

29. Secondary Outcome: Participant Perception of Drug-Free Interval: Duration
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). After the drug-free interval participants were asked, "How would you assess the length of the current drug-free interval?" Participants responded on a scale of 1 (too long) to 5 (too short). Results are reported for participant's perception of the duration of drug-free interval.
Time Frame: Before Cycle 2, 3, 4, 5, 6
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 104
units on a scale
  Before Cycle 2 (n=104) | 2.5 (1.1)
  Before Cycle 3 (n=35) | 2.9 (1.2)
  Before Cycle 4 (n=5) | 1.0 (0.0)
  Before Cycle 5 (n=1) | 2.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6 (n=1) | 2.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.

30. Secondary Outcome: Participant Perception of Drug-Free Interval: Relapse of Symptoms
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). Before the drug-free interval participants were asked, "How much are you concerned about a relapse of symptoms?" After the drug-free interval participants were asked, "Were you concerned about a relapse of symptoms during the drug-free interval?" Participants responded on a scale of 1 (not concerned) to 5 (very much concerned). Results are reported for participant's perception of relapse of symptoms.
Time Frame: Before Cycle 2, 3, 4, 5, 6, after Cycle 1, 2, 3, 4, 5
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  After Cycle 1 (n=115) | 4.4 (0.8)
  Before Cycle 2 (n=106) | 4.1 (1.0)
  After Cycle 2 (n=41) | 4.1 (1.0)
  Before Cycle 3 (n=36) | 4.0 (0.9)
  After Cycle 3 (n=7) | 4.9 (0.4)
  Before Cycle 4 (n=5) | 4.2 (1.1)
  After Cycle 4 (n=3) | 4.3 (0.6)
  Before Cycle 5 (n=1) | 4.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  After Cycle 5 (n=1) | 3.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6 (n=1) | 3.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.

31. Secondary Outcome: Participant Perception of Drug-Free Interval: Effective Therapy After Drug-Free Interval
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). Before the drug-free interval participants were asked, "To what extend are you relieved by the fact that there is an effective therapy after the drug-free interval?" After the drug-free interval participants were asked, "To what extend were you relieved by the fact that there is an effective therapy after the drug-free interval?" Participants responded on a scale of 1 (not much relieved) to 5 (very much relieved). Results are reported for participant's perception of effective therapy after drug-free interval.
Time Frame: Before Cycle 2, 3, 4, 5, 6, after Cycle 1, 2, 3, 4, 5
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 114
units on a scale
  After Cycle 1 (n=114) | 4.6 (0.8)
  Before Cycle 2 (n=106) | 4.4 (0.8)
  After Cycle 2 (n=41) | 4.4 (0.9)
  Before Cycle 3 (n=35) | 4.3 (1.1)
  After Cycle 3 (n=6) | 4.7 (0.8)
  Before Cycle 4 (n=5) | 5.0 (0.0)
  After Cycle 4 (n=2) | 2.5 (2.1)
  Before Cycle 5 (n=1) | 5.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  After Cycle 5 (n=1) | 5.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6 (n=1) | 2.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.

32. Secondary Outcome: Participant Perception of Drug-Free Interval: Disease Activity
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). After the drug-free interval participants were asked, "How would you assess the activity of your disease during the first half of the drug-free interval?" and "How would you assess the activity of your disease during the second half of the drug-free interval?" Participants responded on a scale of 1 (no activity) to 5 (strongest possible activity). Results are reported for participant's perception of disease activity during the first half and second half of drug-free interval.
Time Frame: Before Cycle 2, 3, 4, 5, 6
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 102
units on a scale
  Before Cycle 2-first half (n=102) | 2.4 (1.0)
  Before Cycle 2-second half (n=101) | 3.3 (1.0)
  Before Cycle 3-first half (n=36) | 2.3 (1.0)
  Before Cycle 3-second half (n=36) | 3.0 (1.1)
  Before Cycle 4-first half (n=4) | 2.5 (0.6)
  Before Cycle 4-second half (n=4) | 3.3 (1.3)
  Before Cycle 5-first half (n=1) | 2.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 5-second half (n=1) | 3.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6-first half (n=1) | 1.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6-second half (n=1) | 2.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.

33. Secondary Outcome: Participant Perception of Drug-Free Interval: Satisfaction With Skin Condition
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). After the drug-free interval participants were asked, "How much were you satisfied with the condition of your skin during the first half of the drug-free interval?" and "How much were you satisfied with the condition of your skin during the second half of the drug-free interval?" Participants responded on a scale of 1 (very dissatisfied) to 5 (very satisfied). Results are reported for participant's satisfaction with their skin condition during the first half and second half of drug-free interval.
Time Frame: Before Cycle 2, 3, 4, 5, 6
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 100
units on a scale
  Before Cycle 2-first half (n=100) | 3.3 (1.2)
  Before Cycle 2-second half (n=100) | 2.7 (1.0)
  Before Cycle 3-first half (n=36) | 3.2 (1.4)
  Before Cycle 3-second half (n=36) | 2.8 (1.1)
  Before Cycle 4-first half (n=4) | 3.5 (1.3)
  Before Cycle 4-second half (n=4) | 2.3 (1.0)
  Before Cycle 5-first half (n=1) | 4.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 5-second half (n=1) | 3.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6-first half (n=1) | 4.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6-second half (n=1) | 3.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.

34. Secondary Outcome: Participant Perception of Drug-Free Interval: Risk for Adverse Drug Reactions
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). Before and after the drug-free interval participants were asked to respond on a scale of 1 (no agreement) to 5 (complete agreement) to the statement, "A drug-free interval reduces the risk for adverse drug reactions." Results are reported for participant's perception of risk of adverse drug reactions.
Time Frame: Before Cycle 2, 3, 4, 5, 6, after Cycle 1, 2, 3, 4, 5
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 110
units on a scale
  After Cycle 1 (n=110) | 3.0 (1.1)
  Before Cycle 2 (n=100) | 3.2 (1.3)
  After Cycle 2 (n=41) | 2.9 (1.3)
  Before Cycle 3 (n=38) | 3.1 (1.3)
  After Cycle 3 (n=6) | 2.3 (1.4)
  Before Cycle 4 (n=5) | 1.6 (0.9)
  After Cycle 4 (n=1) | 3.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 5 (n=1) | 3.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  After Cycle 5 (n=1) | 5.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6 (n=1) | 5.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.

35. Secondary Outcome: Participant Perception of Drug-Free Interval: Reminder of Disease
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). Before and after the drug-free interval participants were asked to respond on a scale of 1 (no agreement) to 5 (complete agreement) to the statement, "During drug-free interval I will not be reminded permanently of my disease." Results are reported for participant's perception of reminder of disease during the drug-free interval.
Time Frame: Before Cycle 2, 3, 4, 5, 6, after Cycle 1, 2, 3, 4, 5
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 104
units on a scale
  After Cycle 1 (n=104) | 2.4 (1.3)
  Before Cycle 2 (n=103) | 2.5 (1.3)
  After Cycle 2 (n=39) | 2.7 (1.3)
  Before Cycle 3 (n=38) | 2.7 (1.3)
  After Cycle 3 (n=5) | 1.6 (0.9)
  Before Cycle 4 (n=5) | 1.6 (0.9)
  After Cycle 4 (n=3) | 2.7 (2.1)
  Before Cycle 5 (n=1) | 2.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  After Cycle 5 (n=1) | 5.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6 (n=1) | 5.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.

36. Secondary Outcome: Participant Perception of Drug-Free Interval: Comfort in Everyday Life
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). Before and after the drug-free interval participants were asked to respond on a scale of 1 (no agreement) to 5 (complete agreement) to the statement, "A drug-free interval means more comfort in my everyday life." Results are reported for participant's perception of comfort of life during the drug-free interval.
Time Frame: Before Cycle 2, 3, 4, 5, 6, after Cycle 1, 2, 3, 4, 5
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 104
units on a scale
  After Cycle 1 (n=104) | 2.3 (1.2)
  Before Cycle 2 (n=103) | 2.6 (1.3)
  After Cycle 2 (n=39) | 2.6 (1.3)
  Before Cycle 3 (n=38) | 2.6 (1.3)
  After Cycle 3 (n=5) | 1.8 (1.1)
  Before Cycle 4 (n=5) | 1.8 (0.8)
  After Cycle 4 (n=3) | 1.0 (0.0)
  Before Cycle 5 (n=1) | 2.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  After Cycle 5 (n=1) | 5.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.
  Before Cycle 6 (n=1) | 1.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable at this time point.

37. Secondary Outcome: Participant Perception of Drug-Free Interval: Preference to Continuous Therapy
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). Before and after the drug-free interval participants were asked, "If possible, would you prefer a continuous therapy without drug-free interval?" Participants responded as yes or no to the question. Results are reported for participant's preference towards continuous therapy.
Time Frame: Before Cycle 2, 3, 4, 5, 6, after Cycle 1, 2, 3, 4, 5
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 106
participants
  After Cycle 1- No (n=104) | 9 (1.3)
  After Cycle 1- Yes (n=104) | 95 (1.3)
  Before Cycle 2- No (n=106) | 8 (1.1)
  Before Cycle 2- Yes (n=106) | 98 (0.8)
  After Cycle 2- No (n=40) | 8 (0.0)
  After Cycle 2- Yes (n=40) | 32 (NA)
  Before Cycle 3- No (n=42) | 3 (NA)
  Before Cycle 3- Yes (n=42) | 39 (NA)
  After Cycle 3- No (n=7) | 0
  After Cycle 3- Yes (n=7) | 7
  Before Cycle 4- No (n=6) | 0
  Before Cycle 4- Yes (n=6) | 6
  After Cycle 4- No (n=3) | 1
  After Cycle 4- Yes (n=3) | 2
  Before Cycle 5- No (n=1) | 0
  Before Cycle 5- Yes (n=1) | 1
  After Cycle 5- No (n=1) | 0
  After Cycle 5- Yes (n=1) | 1
  Before Cycle 6- No (n=1) | 0
  Before Cycle 6- Yes (n=1) | 1

38. Secondary Outcome: Participant Perception of Drug-Free Interval: Recommendation of Therapy
Description: A questionnaire was filled in by participants to evaluate their perception of drug-free interval before the start of every drug-free interval (after Cycle 1, 2, 3, 4, 5) and after every drug-free interval (before Cycle 2, 3, 4, 5, 6). Before and after the drug-free interval participants were asked, "Would you recommend therapy with Enbrel to other patients with plaque-psoriasis?" Participants responded as yes or no to the question. Results are reported for participant's likeliness to recommend therapy.
Time Frame: Before Cycle 2, 3, 4, 5, 6, after Cycle 1, 2, 3, 4, 5
Population: Efficacy analysis set. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure; 'n' signifies those participants who were evaluable for this measure at the specified time points. Results are not reported for before Cycle 4, 5, 6, and after Cycle 5 as no participant was evaluable at these time points.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 107
participants
  After Cycle 1- No (n=106) | 0 (1.3)
  After Cycle 1- Yes (n=106) | 106 (1.3)
  Before Cycle 2- No (n=107) | 0 (1.1)
  Before Cycle 2- Yes (n=107) | 107 (0.8)
  After Cycle 2- No (n=40) | 1 (0.0)
  After Cycle 2- Yes (n=40) | 39 (NA)
  Before Cycle 3- No (n=42) | 0 (NA)
  Before Cycle 3- Yes (n=42) | 42 (NA)
  After Cycle 3- No (n=7) | 0
  After Cycle 3- Yes (n=7) | 7
  After Cycle 4- No (n=1) | 0
  After Cycle 4- Yes (n=1) | 1

39. Secondary Outcome: Criteria for Treatment Resumption
Description: Criteria for resumption of therapy for another cycle by the physician were specified after the 5 drug-free intervals as 1) new disease activity (NDA), 2) prevention of deterioration (POD), 3) other reasons (included reasons like end of adverse event, frequent occurrence of adverse event or pre-specified therapy scheme), 4) new disease activity and prevention of deterioration, 5) new disease activity and other reason, 6) prevention of deterioration and other reason, and 7) new disease activity, prevention of deterioration, and other reasons.
Time Frame: Before Cycle 2, 3, 4, 5, 6
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 144
participants
  Before Cycle 2-new disease activity (NDA) (n=144) | 90 (1.3)
  Before Cycle 2- POD (n=144) | 42 (1.3)
  Before Cycle 2- other reason (n=144) | 8 (1.1)
  Before Cycle 2- NDA and POD (n=144) | 4 (0.8)
  Before Cycle 2- NDA and other reason (n=144) | 0 (0.0)
  Before Cycle 2- POD and other reason (n=144) | 0 (NA)
  Before Cycle 2- NDA, POD and other reason (n=144) | 0 (NA)
  Before Cycle 3-NDA (n=43) | 15 (NA)
  Before Cycle 3- POD (n=43) | 25
  Before Cycle 3- other reason (n=43) | 2
  Before Cycle 3- NDA and POD (n=43) | 1
  Before Cycle 3- NDA and other reason (n=43) | 0
  Before Cycle 3- POD and other reason (n=43) | 0
  Before Cycle 3- NDA, POD and other reason (n=43) | 0
  Before Cycle 4- NDA (n=8) | 3
  Before Cycle 4- POD (n=8) | 5
  Before Cycle 4- other reason (n=8) | 0
  Before Cycle 4- NDA and POD (n=8) | 0
  Before Cycle 4- NDA and other reason (n=8) | 0
  Before Cycle 4- POD and other reason (n=8) | 0
  Before Cycle 4-NDA, POD and other reason (n=8) | 0
  Before Cycle 5- NDA (n=3) | 2
  Before Cycle 5- POD (n=3) | 1
  Before Cycle 5- other reason (n=3) | 0
  Before Cycle 5- NDA and POD (n=3) | 0
  Before Cycle 5- NDA and other reason (n=3) | 0
  Before Cycle 5- POD and other reason (n=3) | 0
  Before Cycle 5- NDA, POD and other reason (n=3) | 0
  Before Cycle 6- NDA (n=1) | 1
  Before Cycle 6- POD (n=1) | 0
  Before Cycle 6- other reason (n=1) | 0
  Before Cycle 6- NDA and POD (n=1) | 0
  Before Cycle 6- NDA and other reason (n=1) | 0
  Before Cycle 6- POD and other reason (n=1) | 0
  Before Cycle 6- NDA, POD and other reason (n=1) | 0

40. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) or Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Number of participants with AEs included participants affected with both SAEs and non-SAEs.
Time Frame: Cycle 1 Week 0 up to 30 days after end of study (where end of study was Cycle 6 Week 24)
Population: Safety analysis set included all participants with available post-baseline safety data.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 926
participants
  AEs | 273 (10.6)
  SAEs | 59

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 59/926
Other Adverse Events (participants affected / at risk) | 230/926
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=926)
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Phimosis (Congenital, familial and genetic disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Drowning (General disorders) | 1
Fatigue (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site extravasation (General disorders) | 1
Necrosis (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Erysipelas (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 2
Necrotising fasciitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Abdominal infection (Infections and infestations) | 1
Abscess (Infections and infestations) | 1
Chronic tonsillitis (Infections and infestations) | 1
Muscle abscess (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Accident at work (Injury, poisoning and procedural complications) | 1
Accident (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Tuberculosis serology test positive (Investigations) | 1
Weight decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Sleep disorder (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Scrotal erythema (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Renal transplant (Surgical and medical procedures) | 1
Vascular graft (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Epilepsy (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=926)
Leukopenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
External ear inflammation (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Visual impairment (Eye disorders) | 2
Blepharitis (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 3
Periodontitis (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Salivary gland enlargement (Gastrointestinal disorders) | 1
Condition aggravated (General disorders) | 26
Injection site erythema (General disorders) | 12
Injection site inflammation (General disorders) | 8
Rebound effect (General disorders) | 6
Fatigue (General disorders) | 4
Oedema peripheral (General disorders) | 4
Injection site pruritus (General disorders) | 3
Injection site swelling (General disorders) | 3
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 2
Drug ineffective (General disorders) | 2
Impaired healing (General disorders) | 2
Injection site induration (General disorders) | 2
Injection site reaction (General disorders) | 2
Pyrexia (General disorders) | 2
Application site irritation (General disorders) | 1
Chills (General disorders) | 1
Drug intolerance (General disorders) | 1
Feeling cold (General disorders) | 1
Injection site anaesthesia (General disorders) | 1
Injection site dryness (General disorders) | 1
Injection site nodule (General disorders) | 1
Injection site recall reaction (General disorders) | 1
Injection site warmth (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 26
Infection (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 6
Herpes zoster (Infections and infestations) | 6
Gastrointestinal infection (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 4
Erysipelas (Infections and infestations) | 4
Cystitis (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 3
Anogenital warts (Infections and infestations) | 2
Febrile infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumonia primary atypical (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Abdominal injury (Injury, poisoning and procedural complications) | 1
Accident at home (Injury, poisoning and procedural complications) | 1
Drug exposure before pregnancy (Injury, poisoning and procedural complications) | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 5
Drug exposure via breast milk (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Recall phenomenon (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Anal abscess (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood count abnormal (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 1
Heart rate increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 2
Red blood cell sedimentation rate increased (Investigations) | 1
Liver function test abnormal (Investigations) | 4
Transaminases increased (Investigations) | 2
Tuberculosis test positive (Investigations) | 1
Weight increased (Investigations) | 4
White blood cell count decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Podagra (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Myopathy (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Dysplastic naevus syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Ageusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysaesthesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Trigeminal neuralgia (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 6
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Middle insomnia (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Acne conglobata (Skin and subcutaneous tissue disorders) | 1
Alopecia effluvium (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dermatitis papillaris capillitii (Skin and subcutaneous tissue disorders) | 1
Dermographism (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Photosensitivity allergic reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 23
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Immobile (Social circumstances) | 1
Aortic valve replacement (Surgical and medical procedures) | 1
Cataract operation (Surgical and medical procedures) | 1
Dental operation (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Knee operation (Surgical and medical procedures) | 1
Shoulder operation (Surgical and medical procedures) | 1
Wart excision (Surgical and medical procedures) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 5
Thrombophlebitis (Vascular disorders) | 2
Varicose vein (Vascular disorders) | 2
Injection site extravasation (General disorders) | 2
Influenza (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.